CLINICAL TRIAL: NCT03799744
Title: A Phase I Study to Evaluate the Safety, Tolerability, and Efficacy of VCN-01 in Combination With Durvalumab (MEDI4736) in Subjects With Recurrent/ Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Safety,Tolerability,and Efficacy of VCN-01 With Durvalumab in R/M Head and Neck Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut Català d'Oncologia (Other)
Collaborators: Theriva Biologics SL (Industry); BioClever 2005 S.L. (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ICO-VCN-H&N-2018; 2018-001095-38 (EudraCT Number)
Record Dates: First submitted 2018-11-09; First posted 2019-01-10 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Head and Neck Neoplasms; Carcinoma, Squamous Cell of Head and Neck; Metastasis; Recurrence
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Neoplasm Metastasis; Recurrence | interventions — durvalumab

STUDY DESIGN:
Intervention Model Description: This is a phase I trial, multicenter, open label, and dose escalation study. Patients will be entered at each dose level, according to a planned dose escalation schedule. Absence of unacceptable toxicity at the previous dose is required for entering a patient in the subsequent level.
  The investigational treatment will be a single i.v. VCN-01 dose combined with concomitant i.v. durvalumab (MEDI4736) 1500 mg Q4W (Arm I) or durvalumab starting two weeks after VCN-01 administration, "sequential schedule" (Arm II). Patient recruitment in Arm I and Arm II will be performed in parallel based on slot availability. Only one single dose of VCN-01 will be administered to each patient during the trial. Durvalumab will be administered Q4W until disease progression, unacceptable toxicity, withdrawal of consent, or another discontinuation criterion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VCN-01 and Durvalumab; concomitant. (Experimental): Combination VCN-01 (single iv dose) with Durvalumab, Concomitant schedule; Dose Escalation of VCN-01
  Interventions: Genetic: VCN-01; Biological: Durvalumab
- VCN-01 and Durvalumab; sequential (Experimental): Combination VCN-01 (single iv dose) with Durvalumab, Delayed schedule (14 days); Dose Escalation of VCN-01
  Interventions: Genetic: VCN-01; Biological: Durvalumab

INTERVENTIONS:
Genetic: VCN-01 — Dose level 1: 3.3x10^12 viral particles/patient and Dose level 2: 1x10^13 viral particles/patient
Biological: Durvalumab — Dose: 1500 mg Q4W

SUMMARY:
This is a Phase I Study to Evaluate the Safety, Tolerability, and Efficacy of VCN-01 in Combination With Durvalumab (MEDI4736) in Subjects With Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck.

VCN-01 is a genetically modified oncolytic adenovirus characterized by the presence of four independent genetic modifications on the backbone of the wild-type HAd5 adenovirus genome, encoding human PH20, that confer tumor selectivity and anti-tumor activity.

Durvalumab is a human monoclonal antibody (mAb) of the immunoglobulin G (IgG) 1 kappa subclass that inhibits binding of PD-L1.

The proposed mechanism of action (MOA) for durvalumab is interference in the interaction of PD-L1 with PD-1 and CD80 (B7.1). Blockade of PD-L1/PD-1 and PD-L1/CD80 interactions releases the inhibition of immune responses, including those that may result in tumor elimination.

DETAILED DESCRIPTION:
* Research Hypothesis The presence of VCN-01 into the tumor after systemic administration will help to overcome the observed resistance to durvalumab and other PD1/PD-L1 checkpoint inhibitors.
* Primary objectives To evaluate the safety and tolerability of a single intravenous injection of VCN-01 combined with durvalumab in two administration regimens (concomitant or durvalumab starting two weeks later "sequential schedule"), and to determine the recommended phase II dose (RP2D) of the combination.
* Study design This is a phase I trial, multicenter, open label, and dose escalation study. Patients will be entered at each dose level, according to a planned dose escalation schedule. Absence of unacceptable toxicity at the previous dose is required for entering a patient in the subsequent level.
* Number of Centers: up to 3
* Number of Patients: 15-20 patients
* Study Population: Patients with metastatic squamous cell carcinoma of the head and neck who have progressed during or after treatment with immune-checkpoint inhibitors.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and any locally-required authorization (e.g., Data Privacy Directive in the EU) obtained from the patient prior to performing any protocol-related procedures; including screening evaluations must be obtained.
2. Adult subjects; age ≥ 18 years at time of study entry
3. ECOG Performance status 0 or 1
4. Life expectancy above 3 months
5. Body weight >30kg
6. Adequate normal organ and marrow function as defined below (transfusions intended to elevate any parameters below solely for the intent of meeting study eligibility are not permitted):

   * Leukocytes ≥3000 mcL
   * Absolute neutrophil count ≥1500 mcL (or 1.0) x (≥ 1500 per mm3)
   * Platelets ≥100 000 mcL
   * Haemoglobin ≥9 g/dL
   * Total bilirubin ≤1.5 x ULN; total bilirubin ≤3×ULN in patients with documented Gilbert's Syndrome (unconjugated hyperbilirubinaemia) or in the presence of liver metastases
   * ALT and AST ≤2.5×ULN if no demonstrable liver metastases or ≤5×ULN in the presence of liver metastases
   * Creatinine ≤ 1.5 x UNL or measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance (see section 4.1.).
7. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients (see section 4.1.).
8. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
9. Have histologically and/or cytologically confirmed head and neck squamous cell carcinoma from the specific sites: oral cavity, oropharynx, larynx or hypopharynx that is recurrent/Mestastasic (R/M) and not amenable to curative therapy by surgery or radiation.
10. For patients in R/M disease: has undergone ≥1 previous regimens of cytoreductive chemo-therapies including prior exposure to anti-PD-(L)1. Patients have progressed or be refractory to anti-PD1 or anti-PDL1 therapy. Note: anti-PD1 or Anti-PDL1 therapy with other agents is acceptable. For patients with locally advanced disease those who has progressed in the last 6 months to previous line that include anti-PD1 or anti PD-L1 in the radical treatment.
11. Subjects must have at least 1 lesion that is measurable using RECIST guidelines. RECIST lesions must not have been previously treated with surgery, radiation therapy, or radiofrequency ablation unless there is documented progression after therapy.
12. Subjects must consent to provide paired pretreatment and on-treatment tumor biopsies (1 pre; 2 post).
13. Levels of neutralizing antibodies against adenovirus ≤1/350 dilution
14. All patients are required to have a fibroscan assessment performed during the screening period. Patients with fibrosis value ≥9.5 kPa will not be eligible.

Exclusion Criteria:

1. Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumour embolization, monoclonal antibodies) within 4 weeks (28 days) prior to the first dose of study treatment. Enrolment with a shorter period of time might be allowed upon discussion with the Study Physician/Medical Monitor according data of sufficient washout time form PK properties of the agent.
2. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
3. Previous treatment PD1/PD-L1 inhibition (including Durvalumab) is a specific entry criterion, but patients:Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.

   * All AEs while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study.

     o Exception: Patients with endocrine AE of ≤Grade 2 are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic.
   * Must not have experienced a ≥Grade 3 immune related AE or an immune related neurologic or ocular AE of any grade while receiving prior immunotherapy.
   * Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of > 10 mg prednisone or equivalent per day.
4. Presently has a second malignancy other than SCCHN, or history of treatment for invasive cancer other that SCCHN in the past 3 years except for:

   1. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
   2. Previously treated non-invasive in-situ carcinoma.
   3. Cervical carcinoma stage 1B or less.
   4. Non-invasive basal cell and squamous cell skin carcinoma.
   5. Radically treated prostate cancer (prostatectomy or radiotherapy) with normal prostate-specific antigen, and not requiring ongoing antiandrogen hormonal therapy.
   6. Other malignancy treated with curative intent and with no known active disease ≥3 years before the first dose of study drug and of low potential risk for recurrence.
   7. Patients with other malignancies treated with curative intent and with no known active disease < 3 years and at low risk of recurrence, may be eligible upon discussion with the Medical Monitor.
5. Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Fridericia's Correction (within 15 minutes at 5 minutes apart).
6. Current or prior use of immunosuppressive medication within 28 days before the first dose of VCN-01/durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. Exceptions defined in section 4.2.
7. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values considered not clinically significant or correctable by the investigator. The eligibility of patients who are still experiencing irreversible toxicity that is not reasonably expected to be exacerbated by the study drugs in this study (eg, hearing loss) must be reviewed and approved by the Study Physician. Patients with Grade ≥2 neuropathy or hearing loss will be evaluated on a case-by-case basis after consultation with the Study physician/Medical Monitor.
8. Has experienced immune-related AEs (irAEs) while receiving prior immunotherapy (including anti-CTLA4 treatment) and assessed as CTCAE grade ≥3
9. Has an active or prior documented autoimmune or inflammatory disorder (including but not limited to inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). (See section 4.2 for details and exceptions.)
10. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment.

    Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
11. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug.
12. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent or other minor procedures are acceptable.
13. History of allogenic organ transplantation.
14. Uncontrolled intercurrent illness, including but not limited to, uncontrolled ongoing or active infection (including viral emergent infections), symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent. Exception: patients who are finalizing their antibiotic treatment (for example 3 days left of a total of 7 or 10) for a respiratory tract infection are allowed to be included.
15. History of leptomeningeal carcinomatosis
16. Has untreated central nervous system (CNS) metastases identified either on the baseline brain imaging obtained during the screening period or identified prior to signing the ICF. Patients whose brain metastases have been treated may participate provided they show radiographic stability (defined as 2 brain images, both of which are obtained after treatment to the brain metastases. These imaging scans should both be obtained at least four weeks apart and show no evidence of intracranial progression). In addition, any neurologic symptoms that developed either as a result of the brain metastases or their treatment must have resolved or be stable either, without the use of steroids, or with stable doses of anticonvulsants and/or steroids. Steroid dose must be ≤10mg/day of prednisone or its equivalent (and anticonvulsants) for at least 14 days prior to the start of treatment.
17. Has a history of primary immunodeficiency
18. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (positive HBV surface antigen (HBsAg) result), hepatitis C (positive HCV RNA), or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBcAb] and absence of HBsAg) are eligible. HBV DNA must be obtained in these patients prior to treatment. HBV carriers of those patients requiring antiviral therapy treatment of hepatitis B virus or Hepatitis C are not eligible to participate. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Patients with past or resolved tuberculosis are eligible.
19. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
20. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control (according to the HMA CTFG guidelance) from screening to 90 days after the last dose of durvalumab.
21. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
22. Viral syndrome diagnosed during the two weeks before inclusion
23. Patients receiving full-dose anticoagulant/antiplatelet therapy.
24. Patients with Li Fraumeni syndrome or with previous known retinoblastoma protein pathway germinal deficiency.
25. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety by means of Adverse Events (AEs) | through study completion, an average of 2 years
  Incidence of Adverse Events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Objective response rate (ORR) | On Cycle 3 (+/- 3 days, each cycle is 28 days), and then every 2 cycles (± 7 days) until disease progression or withdrawal (an average of 2 years)
  Proportion of patients with reduction in tumor burden of a predefined amount assessed by CT or MRI
Progression Free Survival (PFS) | On Cycle 3 (+/- 3 days, each cycle is 28 days), and then every 2 cycles (± 7 days) until disease progression or withdrawal (an average of 2 years)
  Time from study enrollment until disease progression or death assessed by CT or MRI
Maximum Plasma Concentration (Cmax ) of VCN-01 | For both arms: On day 1 pre-dose (within 15 minutes prior to VCN-01 infusion) and then 30 minutes, 1, 2, 4, 6, 24 and 48 hours post VCN-01 administration.
  The maximum (or peak) concentration that VCN-01 achieves in plasma after its administration.
Tmax of VCN-01 | VCN-01 and Durvalumab concomitant arm: On day 1 pre-dose (within 15 minutes prior to VCN-01 infusion) and then 30 minutes, 1 hours, 2 hours, 4 hours, 6 hours, 24 hours and 48 hours post VCN-01 administration. VCN-01 and Durvalumab sequential: On day 1
  Time to Maximum Plasma Concentration of VCN-01
AUC of VCN-01 | VCN-01 and Durvalumab concomitant arm: On day 1 pre-dose (within 15 minutes prior to VCN-01 infusion) and then 30 minutes, 1 hours, 2 hours, 4 hours, 6 hours, 24 hours and 48 hours post VCN-01 administration. VCN-01 and Durvalumab sequential: On day 1
  The definite integral in a plot of drug concentration in blood plasma vs. time.
Apparent Half-Life (t1/2) of VCN-01 | VCN-01 and Durvalumab concomitant arm: On day 1 pre-dose (within 15 minutes prior to VCN-01 infusion) and then 30 minutes, 1 hours, 2 hours, 4 hours, 6 hours, 24 hours and 48 hours post VCN-01 administration. VCN-01 and Durvalumab sequential: On day 1
  The time it takes for half to be removed
Elimination rate constant of VCN-01 | VCN-01 and Durvalumab concomitant arm: On day 1 pre-dose (within 15 minutes prior to VCN-01 infusion) and then 30 minutes, 1 hours, 2 hours, 4 hours, 6 hours, 24 hours and 48 hours post VCN-01 administration. VCN-01 and Durvalumab sequential: On day 1
  The rate at which VCN-01 is removed from the body.
VCN-01 viral shedding in blood | VCN-01 and Durvalumab concomitant arm: On day 1: pre-dose and then, 4 hours, 24 hours and 48 hours post dose, on day 8, day 15, day 22 of cycle 1 (each cycle is 28 days), then on day1 of subsequent durvalumab cycles and at the final visit. Arm II: On day
  Determination of VCN-01 levels in peripheral blood samples
anti-VCN-01 antibodies | At screening, on day 1 pre-dose (within 15 minutes prior to VCN-01 ) in both arms. In concomitant arm: at day1 of subsequent durvalumab cycles (each cycle is 28 days), and at the final visit. In sequential arm: at day15 on cycle 1, at day1 of subsequent
  Assessment of Blood levels of neutralizing anti-VCN-01 antibodies
VCN-01 viral shedding in stool and sputum | VCN-01 and Durvalumab concomitant arm: at day 1, 8, 15 and 22 on cycle 1 (each cycle is 28 days) And at day1 of subsequent durvalumab cycles. VCN-01 and Durvalumab sequential: at day -14, -7, 1, 8, 15 on cycle 1 and at day 1 of subsequent durvalumab
  Determination of VCN-01 levels in stool and sputum
Immunological changes induced by the combination of VCN-01 and durvalumab. | VCN-01 and Durvalumab concomitant arm: On day 1: pre-dose, at 30 minutes, 6 hours, 24 hours, 48 hours, at day 8 on cycle 1 (each cycle is 28 days), at day 1of cycle 2 and at the final visit. VCN-01 and Durvalumab sequential: On day 1, 15 minutes before
  Study of the Immunological changes induced by the combination of VCN-01 and durvalumab by assessment of blood levels of circulating Interleukin 6 and Interleukin 10
Changes in Microbiome in stool (VCN-01 and Durvalumab concomitant arm) | On day 1: pre-dose and 1st deposition after-dose (the first deposition occurred from day 1 to day 7), day 8, day 15, day 22 on cycle 1 (each cycle is 28 days).
  Analyse the microbiome in stool, prior and after VCN-01 administration
Changes in Microbiome in stool (VCN-01 and Durvalumab sequential) | On day -14 (pre-dose and 1st deposition after-dose), day -7, Day 1, day 8 and day15 on cycle 1 (each cycle is 28 days).
  Analyse the microbiome in stool, prior and after VCN-01 administration
Circulating free DNA (cfDNA) in plasma analysis (VCN-01 and Durvalumab concomitant arm) | Pre-dose on day 1 (within 15min prior to VCN-01 infusion) and at day 8 on cycle 1, at day 1 on cycle 2, at day 1 on cycle 3 and at day 1 on cycle 4 (within 15min prior durvalumab administration) (each cycle is 28 days).
  To analyse the circulating free DNA (cfDNA) in plasma obtained from samples collected prior and post VCN-01 treatment.
Circulating free DNA (cfDNA) in plasma analysis (VCN-01 and Durvalumab sequential) | On day -14 pre-dose and 1st deposition after-dose(the first deposition occurred from day -14 to day -8), day -7, day 1, day 8 and day15 on cycle 1 (each cycle is 28 days).
  To analyse the circulating free DNA (cfDNA) in plasma obtained from samples collected prior and post VCN-01 treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Institut Català D'Oncologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona